CLINICAL TRIAL: NCT05868655
Title: The Effect of Exercise on Amateur American Football Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, hazal genc, physiotherapist PhD, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: American Football Players
Record Dates: First submitted 2023-04-17; First posted 2023-05-22 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Athletic Injuries
MeSH Terms: conditions — Athletic Injuries | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Prior to and following the eight-week application, evaluation was conducted.
Who Masked: Investigator
Masking Description: Treatment and assessment in the study was performed by different physiotherapists.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise withVideo-Based (Experimental)
  Interventions: Other: Exercise with Video-Based
- Standart Exercise-Home-Based (Active Comparator)
  Interventions: Other: Standart exercise-Home-Based

INTERVENTIONS:
Other: Exercise with Video-Based — A program of stability and balance exercises will be provided
  Arms: Exercise withVideo-Based
Other: Standart exercise-Home-Based — Participants will be asked to take the final measurements after the exercises have been monitored by a physical therapist for eight weeks.
  Arms: Standart Exercise-Home-Based

SUMMARY:
Football is a team activity that calls for numerous sophisticated talents, including speed, endurance, speed, strength, and quickness. It is getting more and more popular among professional and amateur players, particularly in America.

DETAILED DESCRIPTION:
Current research demonstrates that characteristics of American football players like body composition, sprint performance, metabolism, and strength are influenced by elements like the league played, training history, and position played. The ability to generate power with both the upper and lower bodies, change direction quickly, accelerate quickly in both positive and negative directions, run quickly, engage in high-intensity collisions repeatedly, and maintain muscular strength endurance are all skills that players on the court may need.

ELIGIBILITY:
Inclusion Criteria:

* Male individuals between the ages of 18-25
* Being an American football player
* Regular attendance at training sessions

Exclusion Criteria:

* Known neurological disorder
* Serious orthopedic disorders that will prevent him from exercising
* cognitive impairment

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 43 (Actual)
Dates: Start 2023-04-17 (Actual); Primary Completion 2023-06-17 (Actual); Study Completion 2024-08-17 (Actual)

PRIMARY OUTCOMES:
The Tampa Kinesiophobia Scale | 8 weeks
  The Tampa Kinesiophobia Scale is one of two scales that assesses pain-related fear. This scale, which is frequently used in the literature, is based on avoidance due to fear, fear in work-related activities, fear of movement or re-injury. The Tampa Scale for Kinesiophobia is a 17-item questionnaire that quantifies fear of movement.The original 17-item version of the scale creates scores ranging between 17 and 68 with higher scores indicating more fear of movement
Optojump | 8 weeks
  The system can be activated with 2 cameras and at least 2 Optojump bars. In the measurements, the vertical jump height was recorded with the optoJump system and the software of this system (Microgate, Bolzano, Italy). The measurement of the vertical jump distance in centimeters is done by means of two bars in the OptoJump system with sensors that detect movement.
The duration of the jump (milliseconds) .(Optojump) | 8 weeks
  The system can be activated with 2 cameras and at least 2 Optojump bars. The duration of the jump (milliseconds).
The Biodex balance system | six weeks
  The Biodex balance system (BDS) is one of the mechanical platforms frequently used in balance measurements. It assesses balance through a platform that oscillates in the anteroposterior, mediolateral and general directions simultaneously.

SECONDARY OUTCOMES:
Sit-Reach Test | 8 weeks
  The classical sit-reach test will be used to assess flexibility. According to meta-analyses, the classical sit-reach test is the most reliable method to evaluate hamstring flexibility.

CONTACTS AND LOCATIONS:
Locations (1):
- HAZAL genç, Istanbul, None Selected, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fullagar HHK, McCunn R, Murray A. Updated Review of the Applied Physiology of American College Football: Physical Demands, Strength and Conditioning, Nutrition, and Injury Characteristics of America's Favorite Game. Int J Sports Physiol Perform. 2017 Nov 1;12(10):1396-1403. doi: 10.1123/ijspp.2016-0783. Epub 2017 Dec 19. PMID 28338375